CLINICAL TRIAL: NCT07005986
Title: Role of Circulating Pyrophosphate as a Biomarker of Mediacalcinosis in Type 2 Diabetic Patients
Acronym: PPi-Diab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-AOIP-04; IDRCB (Registry Identifier: 2025-A00626-43)
Record Dates: First submitted 2025-05-19; First posted 2025-06-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Patients
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasmatic PPi level, ENPI level and CT-scan of coronary arteries and lower limbs arteries (Experimental)
  Interventions: Diagnostic Test: Plasmatic PPi level

INTERVENTIONS:
Diagnostic Test: Plasmatic PPi level — Plasmatic PPi level dosage at visit 1

SUMMARY:
Type 2 diabetes currently affects around 4 million people in France, with the number of cases rising steadily. Complications of T2DM are essentially cardiovascular. In particular, T2DM is associated with calcification of peripheral vessel walls (mediacalcosis), responsible for increased vascular stiffness. This calcium deposition is known to be a cardiovascular risk factor, but the mechanism of its deposition in relation to diabetes is not clearly established. An important blood compound, inorganic pyrophosphate (PPi), which is the body's natural anti-calcifier is impacted in some way in T2DM. PPi is degraded by alkaline phosphatase (ALP), and is produced by an enzyme called ENPP1. ENPP1 activity is decreased and APL activity increased in insulin-resistant subjects, which could contribute to a decrease in tissue and circulating PPi, and thus favor a tissue pro-calcifying balance. We propose to test this hypothesis in a pilot study characterizing plasma PPi levels, in relation to ENPP1 activity, in type 2 diabetic patients. The aim of the study is also to determine if there is a link between blood PPi levels and the progression of calcifications in arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men (between 40 and 70 years of age).
2. T2DM defined according to ADA or HAS criteria, evolving for more than 6 months, may be : - Not complicated

   * Complicated by diabetic retinopathy and/or diabetic nephropathy (creatinine clearance > 60 ml/min) and/or peripheral arterial disease and/or ischemic heart disease and/or stroke. - With dyslipidemia (LDLc > 1.90) and/or a history of past or active smoking.
   * Balanced with HbA1c < 8% according to patient's personalized objectives, or unbalanced with HbA1c > 9%.
   * Treated with insulin therapy (single or multi-injections) or not. - Whose treatment includes at least one iSGLT2.
3. Member of 'Sécurité Sociale"

Exclusion Criteria:

1. Patient already included in another study.
2. Patient in a particular situation judged incompatible with the study by the investigator.
3. Patient living in a department other than Alpes-Maritimes or Var.
4. Patient refusing to give consent.
5. Patient deprived of liberty by administrative or judicial decision, under guardianship or curatorship.
6. Patient with decompensated hepatic cirrhosis (Child C and above, score 10 to 15 points).
7. Patients with chronic kidney disease (from stage 3, i.e. GFR < 59 ml/min/1.73 m2).
8. Patient with a recent fracture (within the last 3 months).
9. Patient treated with AVK or biphosphonates.
10. Patient with known, treated osteoporosis.
11. Patient with unsupplemented vitamin D deficiency.
12. Patient with active cancer.
13. Patient with an active inflammatory pathology.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-07-18 (Estimated); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Measurement of plasma inorganic pyrophosphate level | Blood samples are taken during first visit, in the morning, after fasting
  Measurement of plasma inorganic pyrophosphate level in Type 2 diabetes patients and comparaison with a laboratory reference value

SECONDARY OUTCOMES:
Coronary and lower limb calcification score | The Computed tomography scan will be performed within two weeks after fisrt visit
  The coronary and lower limb calcification score will be determined using a non-contrast Computed tomography scan of the coronary arteries and lower limbs

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France, France

IPD SHARING:
Plan to Share IPD: No